CLINICAL TRIAL: NCT04021303
Title: Study of the Initiation of Complementary Feeding With a Whole Grain, Gluten-containing Infant Cereal and PROBIOtics to Evaluate Digestive TOLERAance and Immuno-inflammatory Response at the Intestinal Level.
Brief Title: Whole Grain, Gluten-containing Cereal and PROBIOtics to Evaluate Digestive TOLERAance and Immuno-inflammatory Response
Acronym: PROBIOTOLERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PROBIO-TOLERA
Record Dates: First submitted 2019-07-05; First posted 2019-07-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Disorder; Immunologic Diseases in Children
Keywords: Gluten; Probiotic; Prebiotic
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Cereal (Experimental): Experimental cereal with probiotics, prebiotic fiber and low carbohydrates through all the duration of the study.
  Interventions: Dietary Supplement: Experimental cereal
- Conventional cereal (Active Comparator): Conventional gluten free cereal between 4 and 6 months old, and conventional gluten cereal between 7 and 12 months old.
  Interventions: Dietary Supplement: Conventional cereal

INTERVENTIONS:
Dietary Supplement: Experimental cereal — Cereal containing probiotics, prebiotic fiber and low carbohydrates
  Arms: Experimental Cereal
Dietary Supplement: Conventional cereal — Gluten free conventional cereal (from 4 to 6 months old) and conventional cereal with gluten (from 7 to 12 months old)
  Arms: Conventional cereal

SUMMARY:
This study will assess the development of gastrointestinal health in terms of digestive tolerability and immune-inflammatory response at the intestinal level comparing a conventional gluten-free cereal with a new cereal with prebiotics, probiotics and a very moderate amount of gluten. These are products adapted to infant feeding since 4 Months.

DETAILED DESCRIPTION:
In 2008 the ESPGHAN recommended not to give gluten cereals before 4 months but not after 7 months. Although the introduction of gluten in this window was linked to a posible preventive effect on celiac disease, the truth is that it has not been demonstrated. In any case, high exposures to gluten since the 4 months have been associated with a higher incidence of celiac disease and current recommendations propose moderate and progressive exposure to gluten between 4 and 6 months old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (>37 weeks) vaginal delivery
* Adequate birth weight for gestational age (10-90 percentile)
* Infants with normal growth curve (10-90 percentile)
* Infants who were breastfeeding for at least 4 weeks, and at least half of the takes have been by breastfeeding.
* Infants aged 4 months (+/- 1 week) at the time of study inclusion no longer following breastfeeding, or mixed breastfeeding and if they are breast-feeding, no more than one shot a day.
* Availability to continue throughout the study period.
* Signature of informed consent by partents/guardians.

Exclusion Criteria:

* Infants who were born by cesarean section
* Infants born from preconception obese mothers
* Infants born from diabetic mothers or mothers with gestational diabetes
* Infants with a family history of celiac disease (parents or siblings)
* Infants who have had or have some type of allergic manifestation or allergic pathology
* Infants who have needed antibiotic treatment or have received some type of probiotic (the week before inclusion)
* Infants with malformations, diseases or conditions and physical disabilities that cause changes in growth and/or nutritional status
* Infants diagnosed with any immune system-related disease (primary immunodeficiency)
* Infants with a known allergy and/or intolerance to cow's milk protein
* Parents' inability to follow study (at the discretion of the researcher)

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Digestive tolerance | From 4 to 12 months old
  Infant Gastrointestinal Symptom Questionnaire (IGSQ) developed by Riley et al. to be completed by parents/guardians. It contains 13 ítems.For each item there are 5 possible answers in gradation 1 to 5 points and the result is the sum of all of them with minimum scores of 13 (maximum health status) and maximum of 65

SECONDARY OUTCOMES:
Assessing infant feeding habits | At 4, 5, 6, 9 and 12 months old
  Analysis of daily intake through a record of food consumption for 24 hours
Infant microbiota study | Stool sample collected at 4, 6 and 12 months old.
  Composition, diversity of microbiota. This procedure will be performed by studying samples of feces.
Assessment of intestinal health | Stool sample collected at 4, 6 and 12 months old.
  Fecal microbiota profile (fecal pH, butyrate, propionate and acetate) determination
Assessment of immune-inflammatory response | At 4, 6 and 12 months old.
  Record of the IgA secreted in saliva
Infant infection episodes | At 4, 5, 6, 9 and 12 months old.
  Specific parent-reported infant symptoms of mild respiratory, gastrointestinal, skin and oropharyngeal infections. Parents will have a dairy to report all symptoms.
Assessment of infant growth: weight | At 4, 5, 6, 9 and 12 months old.
  Weight measurements in grams to report anthropometric measures
Assessment of infant growth: lenght | At 4, 5, 6, 9 and 12 months old.
  Lenght measurements in centimeters to report anthropometric measures
Assessment of infant growth: cephalic perimeter | At 4, 5, 6, 9 and 12 months old.
  Cephalic perimeter measurements in centimeters to report anthropometric measures
Evolution of body composition | At 4, 5, 6, 9 and 12 months old
  Anthropometric measures (brachial perimeter (mm), trichital skin folds and sub-scapular (mm) with compass lipometer)
Medical history | At 4 months old
  Register of: gestational age, anthropometric measures at birth, lactation data and clinical history of interest
Demographics | At 4 months old
  Parents' age, parent education level, habits and parents lifestyle, home and social environment

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Campoy, Professor, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Medicina, Granada, Spain